CLINICAL TRIAL: NCT04956081
Title: Virtual Neuro-Navigation System for Personalized Community Based TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soterix Medical (Industry)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SMICU061621
Record Dates: First submitted 2021-06-16; First posted 2021-07-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Phase I open-label, 20 subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- virtual neuro-navigation (Experimental): The specific area within the L-DLPFC will be identified by a software using MR images. TMS will be administered to the identified area.
  Interventions: Device: Neuro-navigated Transcranial Magnetic Stimulation (TMS)
- on-line neuro-navigation (Experimental): The specific area within the L-DLPFC will be identified by a person using MR images. TMS will be administered to the identified area.
  Interventions: Device: Neuro-navigated Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Neuro-navigated Transcranial Magnetic Stimulation (TMS) — TMS delivered to a target within the left- dorsolateral prefrontal cortex (L-DLPFC)
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
Phase I study of a virtual neuro-navigation package with built-in support for identifying specific "surface-based" targets to optimze TMS treatment.

DETAILED DESCRIPTION:
Background: Personalized MR neuro-navigation-based targeting approaches have been developed that have the potential to greatly increase TMS efficacy. Nevertheless, these have yet to be incorporated into routine clinical practice because of issues related to 1) the feasibility of neuro-navigation when applied to routine clinical practice, and 2) lack of biomarker-based validation of the critical target across individuals. Recent research at CU has begun to address both feasibility and targeting issues. In the MR-guided neuro-navigation approach, either structural or functional brain scans are used to identify a specific region of interest and the neuro-navigation system is then used to position the TMS coil to target that specific region across individuals. While this approach can be applied within specialized treatment settings, use of these devices requires expertise in 3D brain reconstruction that the majority of TMS providers do not possess. At CU, an initiative is underway to develop a "virtual neuro-navigation" system in which MRI images of the head and brain are uploaded into a server and neuro-navigation is performed "in silico" rather than in person. Scalp coordinates are then relayed to the clinician.

Study: Under this phase I study, Soterix Medical would develop an initial version of the software ("TMSMap") and CU would perform feasibility testing on patients with treatment resistant depression

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of major depressive disorder confirmed using the Mini International Neuropsychiatric Interview (MINI30) Axis 1 and mood modules
* Met criteria for treatment-resistant MDD during the current major depressive episode documented in the MGH Antidepressant Treatment History Questionnaire (ATRQ31), which will be defined as being non-responders (less than 50% of symptom improvement) to two or more depression treatment trials of adequate dose and duration as defined by the MGH ATRQ, as well as an adequate course of TMS treatment using standard targeting approaches (e.g. 5-cm, 5.5-cm, F3)
* at least moderate depression severity, operationalized as Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 20

Exclusion Criteria:

* Ever met criteria for a psychotic disorder (Sz, SzAff, Bipolar disorder), anorexia nervosa or bulimia nervosa within the last year
* Unstable medical condition by history, physical exam or laboratory results
* Currently pregnant or breastfeeding women; fecund women not using adequate contraceptive methods or with plan to become pregnant
* Contraindications to MRI (based on metal screening form)
* Meets criteria for claustrophobia
* Recent drug or alcohol use disorder with DSM-5 specifier of moderate or severe within 6 months, or mild within 2 months; lifetime history of IV drug use
* Actively suicidal, as defined by expressive ideation with a plan or with suicidal ideation that requires immediate medical or treatment intervention.
* A neurological or neuromuscular disorder
* Requires medications for a general medical condition that contraindicate the TMS treatment
* Prior non-response to ECT, vagal nerve stimulation (VNS) or deep brain stimulation (DBS)
* History of ketamine treatment within 6 mo
* History of monoamine oxidase inhibitor (MAOI) within the past month
* Lacks capacity to consent
* Taking medications that increase the risk of seizures.
* For patients on permitted concomitant psychotropic agents (antidepressants, anticonvulsants, benzodiazepines, hypnotics, opiates, triiodothyronine (T3), modafinil, psychostimulants, buspirone, melatonin, omega-3 fatty acids, folate, l-methylfolate, s-adenosyl methionine, lithium) dosing must be stable for at least four weeks prior to study entry and patients must agree to continue at the same dose during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 2 times per week from Baseline until Week 6
  Depression severity scale where higher score indicates greater severity of symptoms

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale Anxiety Somatization Subscale (HAMD-AS)33 | Baseline and at Week 6
  six-item subscale of psychiatric disorder severity where higher score indicates greater severity of symptoms
Side-effect form (SEF) | 2 times per week from Baseline until Week 6
  clinician-rated simple form to document the onset, course, severity, and causality of adverse events
Columbia suicide severity rating scale (C-SSRS) | 2 times per week from Baseline until Week 6
  FDA approved scale for assessment of suicidality
Concomitant Medication List (CML) | 2 times per week from Baseline until Week 6
  This instrument will collect information on all concomitant medications

CONTACTS AND LOCATIONS:
Locations (1):
- Soterix Medical, Inc., Woodbridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No